CLINICAL TRIAL: NCT01544816
Title: Evaluating the Effects of Snack Products on Energy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Cognitive Research Corporation (Industry); Mercer University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KFG-123X-01
Record Dates: First submitted 2012-02-24; First posted 2012-03-06 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Energy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Food Product (Placebo Comparator): Control food product
  Interventions: Other: Snack Product
- Experimental Food Product 1 (Experimental): Experimental food product 1
  Interventions: Other: Snack Product
- Experimental Food Product 2 (Experimental): Experimental food product 2
  Interventions: Other: Snack Product

INTERVENTIONS:
Other: Snack Product — control food product
  Arms: Control Food Product
Other: Snack Product — Experimental food product containing ingredient 1
  Arms: Experimental Food Product 1
Other: Snack Product — Experimental food product containing ingredient 2
  Arms: Experimental Food Product 2

SUMMARY:
To determine the effect of snack products varying in composition, on energy in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must provide informed consent.
2. The subject is male or female, and between the ages of 20 and 45, inclusive.
3. The subject is a routine, moderate daily user of caffeine (approximately 1-4 cups of coffee or equivalent).
4. The subject is fluent in English.
5. The subject has a minimum of a high school diploma.
6. Females of Child-bearing Potential (FOCP) must have a negative urine or serum beta HCG pregnancy test at screening. FOCP must abstain from sexual activity that could result in a pregnancy, or use acceptable contraceptives throughout the period of study treatment exposure. Acceptable contraceptives include IUDs, hormonal contraceptives (oral, implanted or injectable) and double barrier methods (such as condom or diaphragm with spermicidal gel). If hormonal contraceptives are used, the period of use must be sufficiently long to achieve pharmacological effectiveness prior to study treatment exposure (refer to individual product information for details on onset of effectiveness). FOCP who are not currently sexually active, must agree to use acceptable contraception, as defined above, if they decide to become sexually active during the period of study treatment exposure .
7. The subject is in good physical and mental health based on a general medical history.
8. The subject has adequate visual and auditory acuity and cognitive ability to complete the assessments and is capable of understanding and following instructions for the performance tests within the normal, age-adjusted range (within one SD) at screening.
9. Must be able and willing to obtain a minimum of 7 hours of sleep the night prior to each study visit.
10. The subject is willing and able to comply with all requirements defined within this protocol.
11. The subject reports having a snack at least two afternoons per week.
12. The subject reports experiencing an "afternoon slump".

Exclusion Criteria

1. The subject has a current Axis I or Axis II comorbid psychiatric diagnosis or other symptomatic manifestations that, in the opinion of the examining physician (Investigator), will contraindicate treatment with caffeine.
2. Attention Deficit Disorder or Attention Deficit Hyperactivity Disorder
3. BMI ≤ 19 or ≥ 30 kg/m2.
4. The subject has documented allergies, adverse reactions, or intolerance to caffeine.
5. The subject has any significant medical illness or condition for which caffeine is contraindicated.
6. The subject has a history of drug dependence or substance use disorder based upon DSM-IV-TR criteria (excluding nicotine).
7. The subject has a positive urine drug or alcohol drug test result (to include nicotine).
8. The subject has participated in an investigational study or received an investigational drug within the past 28 days.
9. The subject has used nicotine products within 30 days of screening or during the duration of the study.
10. The subject is taking medications, that have CNS effects or affect performance, (such as sedating antihistamines and decongestant sympathomimetics, either oral or topical), and may interfere with efficacy or safety assessments.
11. The subject has a concurrent chronic or acute illness (such as allergic rhinitis or severe cold), disability, or other condition that might confound the results of rating tests administered in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional conditions that, in the Investigator's opinion, would preclude the subject from completing the study or would not be in the best interest of the subject. This would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol.
12. The female subject is pregnant or lactating or planning on becoming pregnant during the study
13. Hypertension or other chronic medical conditions
14. Individuals who do not maintain a routine nighttime sleep schedule (e.g. no shift work).
15. Individuals judged by the Investigator to be unsuitable for enrollment in this study for any reason.
16. The subject has been diagnosed with phenylketonuria.
17. Inability to perform performance tests within the Normal range (i.e., performance no lower than 1SD below the mean) at screening.
18. The subject has a pre-existing medical condition.
19. Subject has been diagnosed with a sleeping disorder.
20. Subject has a fasting glucose of >110 mg/dl.
21. Subject has an allergy to wheat, soy, nuts or other food.
22. Subject has Kosher or Halal dietary restrictions.
23. Subject reports never eating biscuits, cookies or crackers.
24. Epworth Sleepiness Scale ≥ at screening (i.e., evidence of excessive daytime sleepiness).
25. Dislike of chocolate flavorings

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Energy questionnaire OR Rating of perceived energy OR Subjective feeling of energy (visual analog scale) | 90 minutes post snack

CONTACTS AND LOCATIONS:
Overall Officials: Chad VanDenBerg, Pharm.D., Principal Investigator — Mercer University
Locations (1):
- Mercer University Center for Clinical Research, Atlanta, Georgia, United States